CLINICAL TRIAL: NCT03926065
Title: Lunchtime Meal Feeding Study for Preschool Children
Brief Title: Variations in Palatability and Portion Size of Vegetables on Meal Intake of Preschool Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Penn State University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Barbara J. Rolls, Professor of Nutrition and Director of the Laboratory for the Study Human Ingestive Behavior, Penn State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: ChildFood402; R01DK082580 (NIH)
Record Dates: First submitted 2019-04-19; First posted 2019-04-24 (Actual); Results first posted 2020-09-04 (Actual); Last update posted 2020-09-25 (Actual); Status verified 2020-09

CONDITIONS: Feeding Behavior
MeSH Terms: conditions — Feeding Behavior | interventions — Portion Size

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard Palatability and Standard Portion Size (Experimental): Vegetables with Standard Palatability and Standard Portion Size
  Interventions: Other: Plain Vegetables Served in 100% Portion Size
- Standard Palatability and Larger Portion Size (Experimental): Vegetables with Standard Palatability and Larger Portion Size
  Interventions: Other: Plain Vegetables Served in 200% Portion Size
- Enhanced Palatability and Standard Portion Size (Experimental): Vegetables with Enhanced Palatability and Standard Portion Size
  Interventions: Other: Enhanced Vegetables Served in 100% Portion Size
- Enhanced Palatability and Larger Portion Size (Experimental): Vegetables with Enhanced Palatability and Larger Portion Size
  Interventions: Other: Enhanced Vegetables Served in 200% Portion Size

INTERVENTIONS:
Other: Plain Vegetables Served in 100% Portion Size — Lunch includes (a) vegetables without added flavoring (b) the baseline portion size of vegetables
  Arms: Standard Palatability and Standard Portion Size
Other: Plain Vegetables Served in 200% Portion Size — Lunch includes (a) vegetables without added flavoring (b) 200% of the baseline portion size of vegetables
  Arms: Standard Palatability and Larger Portion Size
Other: Enhanced Vegetables Served in 100% Portion Size — Lunch includes (a) vegetables with added flavoring (b) the baseline portion size of vegetables
  Arms: Enhanced Palatability and Standard Portion Size
Other: Enhanced Vegetables Served in 200% Portion Size — Lunch includes (a) vegetables with added flavoring (b) 200% of the baseline portion size of vegetables
  Arms: Enhanced Palatability and Larger Portion Size

SUMMARY:
The aim of the study is to determine the effect of varying both the palatability and portion size of vegetables served to preschool children at a meal on the outcomes of food and energy intake at the meal.

ELIGIBILITY:
Inclusion Criteria:

* Children who are enrolled in a scheduled classroom of the designated childcare centers

Exclusion Criteria:

* Children who are allergic to any of the foods served
* Children whose diets exclude any of the foods served
* Children who will not be present at the childcare center for all of the scheduled study days

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 67 (Actual)
Dates: Start 2019-05-28 (Actual); Primary Completion 2019-10-24 (Actual); Study Completion 2019-10-29 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Laboratory for the Study of Human Ingestive Behavior, The Pennsylvania State University, University Park, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Diktas HE, Roe LS, Keller KL, Sanchez CE, Rolls BJ. Promoting vegetable intake in preschool children: Independent and combined effects of portion size and flavor enhancement. Appetite. 2021 Sep 1;164:105250. doi: 10.1016/j.appet.2021.105250. Epub 2021 Apr 6. PMID 33836215

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Children aged 3 to 5 years old were recruited from classrooms at three childcare centers in State College, Pennsylvania by distributing letters to parents between May 2019 and October 2019.
Groups:
- St Pal/Lg PS, En Pal/St PS, St Pal/St PS, En Pal/Lg PS: Participants who received the meals in the order of Plain Vegetables served in 200% Portion Size first, then Enhanced Vegetables served in 100% Portion Size, then Plain Vegetables served in 100% Portion Size, then Enhanced Vegetables served in 200% Portion Size
- En Pal/Lg PS, St Pal/St PS, En Pal/St PS, St Pal/Lg PS: Participants who received the meals in the order of Enhanced Vegetables served in 200% Portion Size first, then Plain Vegetables served in 100% Portion Size, then Enhanced Vegetables served in 100% Portion Size, then Plain Vegetables served in 200% Portion Size
- En Pal/St PS, En Pal/Lg PS, St Pal/Lg PS, St Pal/St PS: Participants who received the meals in the order of Enhanced Vegetables served in 100% Portion Size first, then Enhanced Vegetables served in 200% Portion Size, then Plain Vegetables served in 200% Portion Size, then Plain Vegetables served in 100% Portion Size
- St Pal/St PS, St Pal/Lg PS, En Pal/Lg PS, En Pal/St PS: Participants who received the meals in the order of Plain Vegetables served in 100% Portion Size first, then Plain Vegetables served in 200% Portion Size, then Enhanced Vegetables served in 200% Portion Size, then Enhanced Vegetables served in 100% Portion Size
- En Pal/Lg PS, St Pal/Lg PS, En Pal/St PS, St Pal/St PS: Participants who received the meals in the order of Enhanced Vegetables served in 200% Portion Size first, then Plain Vegetables served in 200% Portion Size, then Enhanced Vegetables served in 100% Portion Size, then Plain Vegetables served in 100% Portion Size
Period: Study Week 1
Arm/Group | St Pal/Lg PS, En Pal/St PS, St Pal/St PS, En Pal/Lg PS | En Pal/Lg PS, St Pal/St PS, En Pal/St PS, St Pal/Lg PS | En Pal/St PS, En Pal/Lg PS, St Pal/Lg PS, St Pal/St PS | St Pal/St PS, St Pal/Lg PS, En Pal/Lg PS, En Pal/St PS | En Pal/Lg PS, St Pal/Lg PS, En Pal/St PS, St Pal/St PS
Started | 11 | 9 | 14 | 18 | 15
Completed | 11 | 9 | 14 | 18 | 15
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Study Week 2
Arm/Group | St Pal/Lg PS, En Pal/St PS, St Pal/St PS, En Pal/Lg PS | En Pal/Lg PS, St Pal/St PS, En Pal/St PS, St Pal/Lg PS | En Pal/St PS, En Pal/Lg PS, St Pal/Lg PS, St Pal/St PS | St Pal/St PS, St Pal/Lg PS, En Pal/Lg PS, En Pal/St PS | En Pal/Lg PS, St Pal/Lg PS, En Pal/St PS, St Pal/St PS
Started | 11 | 9 | 14 | 18 | 15
Completed | 11 | 9 | 14 | 18 | 15
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Study Week 3
Arm/Group | St Pal/Lg PS, En Pal/St PS, St Pal/St PS, En Pal/Lg PS | En Pal/Lg PS, St Pal/St PS, En Pal/St PS, St Pal/Lg PS | En Pal/St PS, En Pal/Lg PS, St Pal/Lg PS, St Pal/St PS | St Pal/St PS, St Pal/Lg PS, En Pal/Lg PS, En Pal/St PS | En Pal/Lg PS, St Pal/Lg PS, En Pal/St PS, St Pal/St PS
Started | 11 | 9 | 14 | 18 | 15
Completed | 11 | 9 | 14 | 18 | 15
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Study Week 4
Arm/Group | St Pal/Lg PS, En Pal/St PS, St Pal/St PS, En Pal/Lg PS | En Pal/Lg PS, St Pal/St PS, En Pal/St PS, St Pal/Lg PS | En Pal/St PS, En Pal/Lg PS, St Pal/Lg PS, St Pal/St PS | St Pal/St PS, St Pal/Lg PS, En Pal/Lg PS, En Pal/St PS | En Pal/Lg PS, St Pal/Lg PS, En Pal/St PS, St Pal/St PS
Started | 11 | 9 | 14 | 18 | 15
Completed | 11 | 9 | 14 | 18 | 15
Not Completed | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Enrolled participants who completed the study
Arm/Group | Entire Study Population
Number analyzed (Participants) | 67
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.2 (0.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41
  Male | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7
  Not Hispanic or Latino | 59
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 51
  More than one race | 7
  Unknown or Not Reported | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 67

OUTCOME MEASURES:

1. Primary Outcome: Difference Between Interventions in Vegetable Intake
Description: Weight of vegetables consumed at the meal (grams)
Time Frame: One meal per week for each intervention (Study weeks 1, 2, 3, and 4)
Measure: Mean (Standard Error); unit: grams
Arm/Group | Standard Palatability and Standard Portion Size | Standard Palatability and Larger Portion Size | Enhanced Palatability and Standard Portion Size | Enhanced Palatability and Larger Portion Size
Number analyzed (Participants) | 67 | 67 | 67 | 67
grams | 32 (3) | 57 (5) | 31 (3) | 50 (4)
Statistical Analysis 1: Comparison: Standard Palatability and Standard Portion Size vs Standard Palatability and Larger Portion Size vs Enhanced Palatability and Standard Portion Size vs Enhanced Palatability and Larger Portion Size; Standard Palatability (Standard Portion Size and Larger Portion Size) compared to Enhanced Palatability (Standard Portion Size and Larger Portion Size); Test type: Superiority; p = 0.1260, Mixed Models Analysis
Statistical Analysis 2: Comparison: Standard Palatability and Standard Portion Size vs Standard Palatability and Larger Portion Size vs Enhanced Palatability and Standard Portion Size vs Enhanced Palatability and Larger Portion Size; Standard Portion Size (Standard Palatability and Enhanced Palatability) compared to Larger Portion Size (Standard Palatability and Enhanced Palatability); Test type: Superiority; p < 0.0001, Mixed Models Analysis
Statistical Analysis 3: Comparison: Standard Palatability and Standard Portion Size vs Standard Palatability and Larger Portion Size vs Enhanced Palatability and Standard Portion Size vs Enhanced Palatability and Larger Portion Size; Interaction between Portion Size and Palatability; Test type: Superiority; p = 0.0992, Mixed Models Analysis

2. Secondary Outcome: Difference Between Interventions in Food Intake
Description: Weight of food (including milk) consumed at the meal (grams)
Time Frame: One meal per week for each intervention (Study weeks 1, 2, 3, and 4)
Measure: Mean (Standard Error); unit: grams
Arm/Group | Standard Palatability and Standard Portion Size | Standard Palatability and Larger Portion Size | Enhanced Palatability and Standard Portion Size | Enhanced Palatability and Larger Portion Size
Number analyzed (Participants) | 67 | 67 | 67 | 67
grams | 283 (10) | 302 (12) | 287 (10) | 305 (12)
Statistical Analysis 1: Comparison: Standard Palatability and Standard Portion Size vs Standard Palatability and Larger Portion Size vs Enhanced Palatability and Standard Portion Size vs Enhanced Palatability and Larger Portion Size; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.5502, Mixed Models Analysis
Statistical Analysis 2: Comparison: Standard Palatability and Standard Portion Size vs Standard Palatability and Larger Portion Size vs Enhanced Palatability and Standard Portion Size vs Enhanced Palatability and Larger Portion Size; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.0072, Mixed Models Analysis

3. Secondary Outcome: Difference Between Interventions in Meal Energy Intake
Description: Energy consumed at the meal (kilocalories)
Time Frame: One meal per week for each intervention (Study weeks 1, 2, 3, and 4)
Measure: Mean (Standard Error); unit: kilocalories
Arm/Group | Standard Palatability and Standard Portion Size | Standard Palatability and Larger Portion Size | Enhanced Palatability and Standard Portion Size | Enhanced Palatability and Larger Portion Size
Number analyzed (Participants) | 67 | 67 | 67 | 67
kilocalories | 262 (10) | 282 (10) | 277 (8) | 284 (11)
Statistical Analysis 1: Comparison: Standard Palatability and Standard Portion Size vs Standard Palatability and Larger Portion Size vs Enhanced Palatability and Standard Portion Size vs Enhanced Palatability and Larger Portion Size; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.1030, Mixed Models Analysis
Statistical Analysis 2: Comparison: Standard Palatability and Standard Portion Size vs Standard Palatability and Larger Portion Size vs Enhanced Palatability and Standard Portion Size vs Enhanced Palatability and Larger Portion Size; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.0178, Mixed Models Analysis
Statistical Analysis 3: Comparison: Standard Palatability and Standard Portion Size vs Standard Palatability and Larger Portion Size vs Enhanced Palatability and Standard Portion Size vs Enhanced Palatability and Larger Portion Size; Interaction between Portion Size and Palatability; Test type: Superiority; p = 0.2410, Mixed Models Analysis

4. Secondary Outcome: Difference Between Interventions in Meal Energy Density
Description: Energy density of the food consumed at the meal (kilocalories/gram)
Time Frame: One meal per week for each intervention (Study weeks 1, 2, 3, and 4)
Measure: Mean (Standard Error); unit: kilocalories/gram
Arm/Group | Standard Palatability and Standard Portion Size | Standard Palatability and Larger Portion Size | Enhanced Palatability and Standard Portion Size | Enhanced Palatability and Larger Portion Size
Number analyzed (Participants) | 67 | 67 | 67 | 67
kilocalories/gram | 1.41 (0.03) | 1.35 (0.03) | 1.48 (0.03) | 1.40 (0.03)
Statistical Analysis 1: Comparison: Standard Palatability and Standard Portion Size vs Standard Palatability and Larger Portion Size vs Enhanced Palatability and Standard Portion Size vs Enhanced Palatability and Larger Portion Size; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0012, Mixed Models Analysis
Statistical Analysis 2: Comparison: Standard Palatability and Standard Portion Size vs Standard Palatability and Larger Portion Size vs Enhanced Palatability and Standard Portion Size vs Enhanced Palatability and Larger Portion Size; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p < 0.0001, Mixed Models Analysis

5. Other Pre Specified Outcome: Preference of Vegetables Served at the Meal
Description: Preferred version of vegetables (1=standard palatability, 2=enhanced palatability)
Time Frame: Study week 5
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Liking of All Foods Served at the Meal
Description: The Yummy-Yucky Cartoon Faces Scale (1=Yucky, 2=Just Okay, and 3=Yummy)
Time Frame: Study week 5
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Ranking of All Foods Served at the Meal
Description: Ranking of all foods in order of preference (1= most preferred, 2= next most preferred, etc.)
Time Frame: Study week 5
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 5 weeks
Arm/Group | Standard Palatability and Standard Portion Size | Standard Palatability and Larger Portion Size | Enhanced Palatability and Standard Portion Size | Enhanced Palatability and Larger Portion Size
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/67 | 0/67 | 0/67
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/67 | 0/67 | 0/67
Other Adverse Events (participants affected / at risk) | 0/67 | 0/67 | 0/67 | 0/67

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-02-26): https://cdn.clinicaltrials.gov/large-docs/65/NCT03926065/Prot_SAP_000.pdf
  • Informed Consent Form (2020-02-26): https://cdn.clinicaltrials.gov/large-docs/65/NCT03926065/ICF_001.pdf